CLINICAL TRIAL: NCT06428071
Title: Mechanical Knee Decompression With and Without Heating: Impact on Pain, Function, and Range of Motion
Brief Title: Decompression Versus Heat and Decompression in Knee OA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hail (Other)
Responsible Party: Principal Investigator, Hisham Mohamed Hussein, principal investigator, University of Hail
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-2024-265
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: 3 arm parallel randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: This study will be double-blinded consequently neither the assessor nor the data analyzer will be aware of the allocation sequence. Each participant will be coded using special numbers that refer to the correct allocation. The interpretation of these code numbers will be kept with the senior author who will not be involved in the treatment or assessment. The therapist will only be allowed to get the code number interpretation after the end of the allocation process and at the beginning of the study. In this study, the participants and the therapist will be blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard physical therapy program (Active Comparator): All Patients in the three groups will receive supervised systematic exercise therapy that was performed effectively in previous work. This program consisted of lower limb static, dynamic, and flexibility exer¬cises that targeted the quadriceps, hamstrings, and gluteus muscles; and core strength training for 20 minutes per day. This program will be applied 3 times per week for 6 weeks
  Interventions: Other: standard physical therapy
- knee Decompression (Experimental): The ACUTRAC AT270 Traction System device will be used for traction. The patient will assume the supine position with the hip of the treated limb in semi-flexion and the ipsilateral knee in 25-30º flexion. 15 minutes of continuous mechanical traction using 20% of the patient's weight will be used. The session will be 15 minutes, once a day, three-times a week for 6 weeks.
  This group will receive decompression and standard physical therapy.
  Interventions: Other: standard physical therapy; Other: knee Decompression
- Decompression plus heating (Experimental): this group will receive the standard physical therapy, the mechanical decompression and superficial heating using heat pad on the knee joint for 20 minutes while the patient receives the decompression session
  Interventions: Other: standard physical therapy; Other: knee Decompression; Other: hot pack

INTERVENTIONS:
Other: standard physical therapy — All Patients in the three groups will receive supervised systematic exercise therapy that was performed effectively in previous work. This program consisted of lower limb static, dynamic, and flexibility exer¬cises that targeted the quadriceps, hamstrings, and gluteus muscles; and core strength training for 20 minutes per day. This program will be applied 3 times per week for 6 weeks to all the participants
  Other Names: routine physical therapy
Other: knee Decompression — continuous mechanical decompression using 20% of the body weight as a traction force for 15 minutes.
  Other Names: knee traction
  Arms: Decompression plus heating; knee Decompression
Other: hot pack — hot pack over the treated knee joint will be applied for 20 minutes. this application will be performed while the patient is receiving the decompression session
  Other Names: superficial heating; moist heat
  Arms: Decompression plus heating

SUMMARY:
a randomized controlled trial tends to compare the effects of adding superficial heating during the application of knee decompression session to the results of decompression alone without heating.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a progressive multifactorial joint disease characterized by chronic pain and functional disability due to the degeneration of the articular cartilage. The knee joint is the most vulnerable joint in the human body and occupies four-fifths of the burden of OA worldwide. Subjects having KOA demonstrate deferent clinical and radiological characteristics such as narrowed joint space, osteophytes around the articular surface, subchondral sclerosis, pain, limited range of motion (ROM), and declined functional status.

Except for the arthroplasty for the severely arthritic knee joint, there is no cure for the degeneration of joint cartilage. Medications, exercises, and physical agents can be used to address the associated pain, muscular tightness, weakness, and physical disability.

Interestingly, previous efforts that applied traction (decompression) on the arthritic knee joint demonstrated favorable results even on the thickness of the articular cartilage. However, these methods were mainly invasive surgical procedures that encountered disadvantages like the risk of infection and prolonged bedridden that might affect the general health of the patients

ELIGIBILITY:
Inclusion Criteria:

* Both sexes
* age between 45 to 60 years.
* Normal and or overweight categories of BMI 19-30 kg/m2
* Unilateral (grade 2 and 3) knee OA according to the Kellgren-Lawrence radiological rating scale

Exclusion Criteria:

* lower limb deformities as genu varum, valgus, flat foot
* leg length discrepancy
* previous trauma and or surgery to the knee joint
* Bone disease
* Inability to refrain from analgesic/anti-inflammatory medications for 6 weeks

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2024-06-15 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
pain intensity | at base line
  Visual Analog Scale (VAS) will be used to assess pain. This scale is proved to be valid and reliable mean of assessing pain. The patient's pain intensity is represented by a point between the extremes of "no pain at all" and "worst pain imaginable." The outcomes range between no pain to sever pain according to the distance in mm measured from the 0 point of the horizontal line.
pain intensity | after the end of the treatment (after 6 weeks)
  Visual Analog Scale (VAS) will be used to assess pain. This scale is proved to be valid and reliable mean of assessing pain. The patient's pain intensity is represented by a point between the extremes of "no pain at all" and "worst pain imaginable." The outcomes range between no pain to sever pain according to the distance in mm measured from the 0 point of the horizontal line.
active knee range of motion | at baseline
  this outcome will be assessed using a vlaid and reliable android-mobile application designed to assess joint range of motion (ROM). The mobile phone will be secured to the lateral aspect of the leg so that the normal extension will be represented as zero on the app screen. The patient will be asked to move the tested knee from the maximum extension to the maximum available flexion. The value of the angle will be recorded. The difference between the extension angle and flexion angle will be calculated.
active knee range of motion | after the end of the treatment (after 6 weeks)
  this outcome will be assessed using a vlaid and reliable android-mobile application designed to assess joint range of motion (ROM). The mobile phone will be secured to the lateral aspect of the leg so that the normal extension will be represented as zero on the app screen. The patient will be asked to move the tested knee from the maximum extension to the maximum available flexion. The value of the angle will be recorded. The difference between the extension angle and flexion angle will be calculated.
function | at baseline
  It is consisted of 24 questions, five related to pain, two related to stiffness and 17 to physical function. Its reliability was proved in previous work.the questions in this scale takes from 0 to 4 points and the total will be calculated. higher scores indicate more disability
function | after the end of the treatment (after 6 weeks)
  It is consisted of 24 questions, five related to pain, two related to stiffness and 17 to physical function. Its reliability was proved in previous work.the questions in this scale takes from 0 to 4 points and the total will be calculated. higher scores indicate more disability

CONTACTS AND LOCATIONS:
Locations (1):
- Hisham Hussein, Hail, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
the data will be available with the senior author up on request